CLINICAL TRIAL: NCT03307447
Title: Secukinumab Therapy for the Treatment of Moderate to Severe Plaque Psoriasis With Response Monitoring Using Optical Coherence Tomography (OCT).
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Narrows Institute for Biomedical Research (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #1617
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-10

CONDITIONS: Psoriasis Vulgaris
Keywords: optical coherence tomography
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Cosentyx (Secukinumab) 300 mg subcutaneous injection at weeks 0, 1, 2, 3 and 4 followed by every 4 weeks until 16 weeks
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300 mg subcutaneous injection
  Other Names: cosentyx

SUMMARY:
This is a phase IV, single-center, open label, single arm study in which a group of 30 subjects with moderate to severe plaque psoriasis will receive secukinumab therapy. Non-invasive imaging with optical coherence tomography (OCT) will be used to monitor the resolution of psoriatic plaques with treatment in comparison to observed clinical improvements. Early subclinical finding will be used to elucidate drug mechanism of action. Assessment will be based on intrasubject comparisons, and all findings will be compared to patients baseline imaging.

DETAILED DESCRIPTION:
Secukinumab, an anti-IL-17A monoclonal antibody, is an effective treatment for moderate to severe plaque psoriasis.While there is an abundance of clinical data in the literature supporting the clinical efficacy of this therapy, there is limited data on early disease clearance and other histologic findings elucidating a drug mechanism of action. Hyper-proliferation of the epidermis and inflammation of dermis seen in psoriasis are thought to be due to persistent T-cell activation and production of several pro-inflammatory cytokines by dermal immune reaction. Therefore, with treatments with immunomodulatory effects, such as Secukinumab, monitoring markers of inflammation, angiogenesis, and collagen synthesis would be useful in establishing mechanism of action. While a skin biopsy can show these findings at one moment in time, it does not allow for repetitive monitoring overtime. The investigators propose the use of non-invasive imaging with Optical Coherence Tomography (OCT) to demonstrate histologic features of plaque psoriasis not clinically evident. Upon completion of the study, the investigators will assess when OCT improvements of psoriasis treatment are detectable and how these findings correlate to observed clinical improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject at least 18 years of age with a diagnosis of moderate to severe chronic plaque psoriasis vulgaris for at least 6 months.
2. Subjects must be candidates for systemic therapy and have at least moderate to severe psoriasis, as defined by the Psoriasis Area and Severity Index (PASI) score: body surface area (BSA) involvement >10% , PASI >12 and/or IGA modified (mod 2011) score of 3 ("moderate") or 4 ("severe"). [2-4]
3. Patients must be naïve to prior biologic treatment
4. Subject is able to provide written informed consent and comply with the requirements of this study protocol.
5. Subjects who are women of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Acceptable methods of birth control include intrauterine device (IUD); oral, transdermal, implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study); tubal ligation; abstinence and barrier methods with spermicide. Otherwise, if not of childbearing potential, subjects must: have a sterile or vasectomized partner; have had a hysterectomy, a bilateral oophorectomy or be clinically diagnosed infertile; or be in a menopausal state for at least a year.
6. Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) negative at the time of screening, or if patient has a history of positive PPD or QuantiFERON, he/she has completed the appropriate prophylaxis.
7. Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination.

Exclusion Criteria:

1. Patients with guttate, erythrodermic, exfoliative, or pustular psoriasis, other skin conditions affecting the treatment area, severe hepatic disorders or severe renal insufficiency
2. Have received systemic psoriasis treatments (such as psoralen and PUVA light therapy, cyclosporine, corticosteroids, methotrexate, retinoids, mycophenolate, hydroxyurea, azathioprine, sirolimus) or phototherapy within the previous 4 weeks; or have had topical therapy within the previous 2 weeks.
3. Have received any biologic agent for the treatment of psoriasis, including etanercept, infliximab or adalimumab, alefacept, ustekinumab, or any other biologic agent
4. Use of other drugs with potential effect on psoriasis, such as beta blockers, antimalarials, angiotensin-converting enzyme inhibitors, and lithium, are allowed, provided that treatment was not initiated and the dosage did not change during the trial.
5. Any subject who is pregnant or refuses to practice an acceptable method of birth control (as stated in inclusion criterion # 4)
6. History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) at screening. Subjects with a positive or indeterminate PPD or QFT test may participate in the study if a full tuberculosis work up (according to local practice/guidelines) is completed within 12 weeks prior to randomization and establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated at least for 4 weeks prior to randomization and the course of prophylaxis is planned to be completed.
7. Active Crohn's disease
8. History of significant allergies or intolerances
9. Imumunocompromised patients, including Subjects with a history of TB, HIV, Hepatitis B or Hepatitis C infections
10. Have had live vaccination within 12 weeks prior to study
11. Have evidence of active infection, such as fever, within 5 days of dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Elucidate drug mechanism of action by monitoring morphologic changes in lesional vs. perilesional psoriatic plaques using optical coherence tomography (OCT). | week 12
  Lesional and peri-lesional skin will be monitored using OCT for improvement from baseline by measuring changes epidermal, dermal and DEJ, as well as changes in vasculature.

SECONDARY OUTCOMES:
Compare timing of subclinical improvement on OCT to the proportion of patients who achieve a reduction in PASI score by at least 75% (PASI 75) and/or score of 0 or 2-point improvement on the IGA (mod 2011) by week 12. | week 12
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) or achieve a score of 0 on IGA, or at least a 2 point improvement, at week 12.
Compare the onset/timing of subclinical improvement on OCT imaging to patients who achieve a 90% or 100% (PASI 90 and PASI 100) improvement from baseline in the PASI | week 16
  a. To compare the onset/timing of subclinical improvement on OCT imaging to patients who achieve a 90% or 100% (PASI 90 and PASI 100) improvement from baseline in the PASI by week 16

CONTACTS AND LOCATIONS:
Locations (1):
- VA NY Harbor Healthcare System, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided